CLINICAL TRIAL: NCT00138749
Title: An 8-Week, Multi-Centre,Randomised Double-Blind, Placebo Controlled, Parallel Group Study To Evaluate The Efficacy,Toleration And Safety Of (+)- [S,S]- Reboxetine In The Treatment Of Stress Urinary Incontinence (SUI) In Women.
Brief Title: An 8 Week Study Looking At The Efficacy, Toleration And Safety Of SS-RBX For Stress Urinary Incontinence.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061023
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

INTERVENTIONS:
Drug: SS-RBX

SUMMARY:
A study designed to assess the efficacy, toleration and safety of SS-RBX for the treatment of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant stress urinary incontinence

Exclusion Criteria:

* History or evidence of any relevant confounding urological or neurological disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402
Dates: Start 2004-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Proof of concept study to assess the efficacy, tolerability and safety of SS-RBX vs. placebo in the treatment of SUI.

SECONDARY OUTCOMES:
To evaluate whether an upward dose adjustment affects the tolerability of SS-RBX.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (87):
- United States (81):
  - Pfizer Investigational Site, Anchorage, Alaska
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Atherton, California
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Laguna Woods, California
  - Pfizer Investigational Site, Murrieta, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Tarzana, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Vista, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Panama City, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Port Richey, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Alpharetta, Georgia
  - Pfizer Investigational Site, Coeur d'Alene, Idaho
  - Pfizer Investigational Site, Arlington Heights, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Melrose Park, Illinois
  - Pfizer Investigational Site, Greenwood, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Greenbelt, Maryland
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Liberty, Missouri
  - Pfizer Investigational Site, North Kansas City, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Edison, New Jersey
  - Pfizer Investigational Site, West Orange, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Burlington, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Concord, North Carolina
  - Pfizer Investigational Site, Fayetteville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Colmar, Pennsylvania
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Sewickley, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Corsicana, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Sandy City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- Canada (6):
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061023&StudyName=An+8+Week+Study+Looking+At+The+Efficacy%2C+Toleration+And+Safety+Of+SS%2DRBX+For+Stress+Urinary+Incontinence%2E